CLINICAL TRIAL: NCT05063539
Title: Assessment of Safety, Tolerability, and Efficacy of LY3372689 in Early Symptomatic Alzheimer's Disease
Brief Title: A Study of LY3372689 to Assess the Safety, Tolerability, and Efficacy in Participants With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18094; I9X-MC-MTAE (Other: Eli Lilly and Company); 2021-000170-29 (EudraCT Number); 2024-512295-36-00 (EU CTIS Number)
Record Dates: First submitted 2021-09-14; First posted 2021-10-01 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Mild Cognitive Impairment; Prodromal Alzheimer's Disease; Tauopathy; Tau; OGA Inhibitor
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Tauopathies; Pick Disease of the Brain

STUDY DESIGN:
Intervention Model Description: Based on a common closed study design. Participants final endpoint time will be between 76-124 weeks.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.75 Milligram (mg) LY3372689 (Experimental): Participants received 0.75 mg LY3372689 administered orally once daily for up to 124 weeks
  Interventions: Drug: LY3372689
- 3 mg LY3372689 (Experimental): Participants received 3 mg LY3372689 administered orally once daily for up to 124 weeks.
  Interventions: Drug: LY3372689
- Placebo (Placebo Comparator): Participants received placebo administered orally once daily for up to 124 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3372689 — given orally
  Arms: 0.75 Milligram (mg) LY3372689
Drug: LY3372689 — given orally
  Arms: 3 mg LY3372689
Drug: Placebo — given orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and effect of study drug LY3372689 in participants with early symptomatic Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria:

* Gradual and progressive change in memory function reported by participants or informants for ≥ 6 months
* MMSE score of 22 to 30 (inclusive) at screening
* CDR global score of 0.5 to 1.0 (inclusive), with a memory box score ≥0.5.
* Meet 18F flortaucipir positron emission tomography (PET) scan (central analysis) criteria
* Have a study partner who will provide written informed consent to participate

Exclusion Criteria:

* Contraindication to MRI or PET scans
* Have known allergies to LY3372689, related compounds, or any components of the formulations

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2025-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (69):
- United States (35):
  - Hope Clinical Research, Inc., Canoga Park, California
  - Neuro-Pain Medical Center, Fresno, California
  - Irvine Clinical Research, Irvine, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - VIN-Julie Schwartzbard, Aventura, Florida
  - Neurology Offices of South Florida, Boca Raton, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - K2 Medical Research, Maitland, Florida
  - ClinCloud - Viera, Melbourne, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - VIN-Andrew Lerman, Miami, Florida
  - IMIC, Inc., Miami, Florida
  - VIN-Victor Faradji, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - VIN- Margarita Almeida El-Ramey, Pembroke Pines, Florida
  - Brain Matters Research, Stuart, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - Boston Center for Memory, Newton, Massachusetts
  - Donald S. Marks M.D., P.C., Plymouth, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - University at Buffalo - UBMD Neurology, Buffalo, New York
  - Abington Neurological Associates, Ltd., Abington, Pennsylvania
  - Keystone Clinical Studies, Plymouth Meeting, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Kerwin Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The Memory Clinic, Bennington, Vermont
- Australia (11):
  - Central Coast Neurosciences Research (Tumbi Umbi), Central Coast, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - HammondCare Greenwich Hospital, Sydney, New South Wales
  - Hornsby Ku-Ring-Gai Hospital, Sydney, New South Wales
  - KARA Institute for Neurological Diseases, Sydney, New South Wales
  - Private Practice - Dr PL Morris, Southport, Queensland
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - NeuroCentrix, Carlton, Victoria
  - Delmont Private Hospital, Glen Iris, Victoria
  - HammondCare, Malvern, Victoria
- Canada (5):
  - Bruyère Research Institute, Ottawa, Ontario
  - Clinique de la Mémoire de l'Outaouais, Ottawa, Ontario
  - Ottawa Memory Clinic, Ottawa, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
- Japan (9):
  - National Center for Geriatrics and Gerontology, Ōbu, Aichi-ken
  - Himeji Central Hospital Affiliated Clinic, Himeji, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Memory Clinic Toride, Toride, Ibaraki
  - Oita University Hospital, Yufu, Oita Prefecture
  - Katayama Medical Clinic, Kurashiki, Okayama-ken
  - Nozomi Memory Clinic, Mitaka-shi, Tokyo
  - Kikukawa Clinic, Nerima City, Tokyo
  - Memory Clinic Ochanomizu, Tokyo
- Poland (9):
  - Nzoz Neuro-Kard Ilkowski i Partnerzy SPL, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne NEUROMED, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Diamond Clinic, Krakow, Lesser Poland Voivodeship
  - Wroclawskie Centrum Alzheimerowskie, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne NeuroProtect, Warsaw, Masovian Voivodeship
  - Podlaskie Centrum Psychogeriatrii, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne SENIOR, Sopot, Pomeranian Voivodeship
  - Centrum Medyczne Euromedis, Szczecin, West Pomeranian Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.vivli.org/

REFERENCES:
- See also: A Study of LY3372689 to Assess the Safety, Tolerability, and Efficacy in Participants With Alzheimer's Disease — https://trials.lillytrialguide.com/en-US/trial/6wDcj33niQMZDbeYm8iDfu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Current results reporting is only for the primary outcome data per Primary Database Lock (July 9, 2024) and final results will be presented at the time of reporting the final results, i.e., no later than May 22, 2026.
Groups:
- 0.75 Milligrams (mg) LY3372689: Participants received 0.75 mg LY3372689 administered orally once daily for up to 124 weeks.
Period: Overall Study
Arm/Group | 0.75 Milligrams (mg) LY3372689 | 3 mg LY3372689 | Placebo
Started | 110 | 109 | 108
Received at Least 1 Dose of Study Drug (Safety Population) | 108 | 110 (One participant randomized to 0.75 mg LY3372689 moved to 3 mg LY3372689) | 108
Completed | 86 | 70 | 89
Not Completed | 24 | 39 | 19
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Death | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 4 | 3 | 1
Not completed — Progressive Disease | 0 | 2 | 0
Not completed — Withdrawal by Subject | 17 | 26 | 14
Not completed — Withdrawal Due To Caregiver Circumstances | 1 | 1 | 0
Not completed — Subject was Randomized in IWRS prior to Realization that Vital signs would be Exclusionary | 1 | 0 | 0
Not completed — Subject no longer Wished to Continue with IP or Follow-up Visits | 0 | 0 | 1
Not completed — Discontinued due to Common Close Design | 0 | 1 | 0
Not completed — Participant not co-operative | 0 | 1 | 0
Not completed — Patient Moving to Different Place from Where it takes 4 hours to Come to Site to Continue | 0 | 0 | 1
Not completed — Caregiver Withdrew Consent due to Participant Moved to Long Term Care Home | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 0.75 mg LY3372689: Participants received 0.75 mg LY3372689 administered orally once daily for up to 124 weeks.
- Total: Total of all reporting groups
Arm/Group | 0.75 mg LY3372689 | 3 mg LY3372689 | Placebo | Total
Number analyzed (Participants) | 110 | 109 | 108 | 327
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (5.40) | 73.4 (5.38) | 73.4 (5.47) | 73.4 (5.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 63 | 68 | 201
  Male | 40 | 46 | 40 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 2 | 10
  Not Hispanic or Latino | 104 | 102 | 102 | 308
  Unknown or Not Reported | 2 | 3 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 12 | 14 | 11 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 3 | 7
  White | 95 | 94 | 94 | 283
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 14 | 8 | 10 | 32
  Canada | 12 | 12 | 10 | 34
  Japan | 11 | 13 | 11 | 35
  Poland | 16 | 21 | 18 | 55
  United States | 57 | 55 | 59 | 171
Baseline Integrated Alzheimer's Disease Rating Scale (iADRS) Score [Mean (Standard Deviation); unit: Score on a scale] — Integrated Alzheimer's Disease Rating Scale is used to assess whether LY3372689 slows down the clinical decline associated with Alzheimer's disease (AD) compared with placebo. iADRS is an integrated assessment of cognition and daily function comprised of items from the Alzheimer's disease assessment scale-cognitive subscale (ADAS-Cog13) and the Alzheimer's disease cooperative study-instrumental activities of daily living scale (ADCS-iADL). The scale ranges from 0 to 144, where lower scores indicate worse performance and higher score indicates better performance
  Score on a scale | 111.8 (11.99) | 109.3 (13.25) | 110.4 (12.77) | 110.5 (12.68)
Screening Tau Category [Count of Participants; unit: Participants] — All randomized participants (pts) who have only evaluable Screening Tau category data. Intermediate tau (Low-medium): All pts with screening composite tau PET standardized uptake value ratio (SUVr) <= 1.46 and a topographic deposition pattern consistent with advanced AD (AD++) or 1.10 <= SUVr <= 1.46 and a topographic deposition pattern consistent with moderate AD (AD+).
  High tau:All pts with SUVr >1.46 and topographic deposition pattern consistent with either moderate (AD+) or advanced AD (AD++).
  Participants
    Intermediate (Low-medium) | 87 | 86 | 86 | 259
    High | 23 | 23 | 22 | 68

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End Time Point in Integrated Alzheimer's Disease Rating Scale (iADRS) (Intermediate (Low-medium) Tau Population)
Description: iADRS is a simple linear combination of scores from 13-item alzheimer's disease assessment scale-cognitive subscale (ADAS-Cog13) and the Alzheimer's disease cooperative study-instrumental activities of daily living scale (ADCS-iADL). It is used to assess whether LY3372689 slows down the cognitive and functional decline associated with early symptomatic Alzheimer's Disease, compared to placebo. The iADRS score ranges from 0 to 144 with lower scores indicating worse performance and higher score better performance. Change from baseline was calculated using Bayesian disease progression model (DPM) adjusted for age at baseline, AChEI/Memantine use at baseline, pooled investigator. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 100
Population: All randomized participants with baseline or post-baseline data for this outcome with baseline Intermediate Tau level.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 0.75 mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 86 | 85 | 84
score on a scale | -8.39 [-10.219 to -6.640] | -13.27 [-15.481 to -11.097] | -10.07 [-11.900 to -8.338]
Statistical Analysis 1: Comparison: 0.75 mg LY3372689 vs Placebo; Test type: Superiority; Posterior Mean Difference = 1.68, 95% CI 2-sided [-0.375 to 3.771] — Posterior mean difference with 95% credible interval is reported
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Test type: Superiority; Posterior Mean Difference = -3.20, 95% CI 2-sided [-5.354 to -1.042] — Posterior mean difference with 95% credible interval is reported

2. Secondary Outcome: Change From Baseline to End Time Point in iADRS (Overall Population)
Description: iADRS is a simple linear combination of scores from 13-item alzheimer's disease assessment scale-cognitive subscale (ADAS-Cog13) and the Alzheimer's disease cooperative study-instrumental activities of daily living scale (ADCS-iADL). It is used to assess whether LY3372689 slows down the cognitive and functional decline associated with early symptomatic Alzheimer's Disease, compared to placebo. The iADRS score ranges from 0 to 144 with lower scores indicating worse performance and higher score better performance. Change from baseline was calculated using Bayesian disease progression model (DPM) adjusted for age at baseline, baseline tau PET category, AChEI/Memantine use at baseline, pooled investigator. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 100
Population: All randomized participants with baseline or post-baseline data for this outcome.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 0.75 mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 109 | 108 | 106
score on a scale | -10.48 [-12.247 to -8.739] | -17.14 [-19.379 to -14.900] | -12.07 [-13.916 to -10.370]
Statistical Analysis 1: Comparison: 0.75 mg LY3372689 vs Placebo; Test type: Superiority; Posterior Mean Difference = 1.59, 95% CI 2-sided [-0.443 to 3.697] — Posterior mean difference with 95% credible interval is reported
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Test type: Superiority; Posterior Mean Difference = -5.07, 95% CI 2-sided [-7.277 to -2.862]

3. Secondary Outcome: Change From Baseline to End Time Point in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) (Intermediate (Low-medium) Tau Population)
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score are assigned for each of 6 domains; Total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity. LS Mean change from baseline was calculated using natural cubic spline with 2 degrees of freedom (NCS2) adjusted for fixed effects of NCS basis expansion terms (two terms), NCS basis expansion term-by-treatment interaction, visit (in weeks), investigator site (pooled), age at baseline, AChEI/Memantine use at baseline.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline or post-baseline data for this outcome with baseline Intermediate Tau level.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- 0.75mg LY3372689: Participants received 0.75 mg LY3372689 administered orally once daily for up to 124 weeks.
Arm/Group | 0.75mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 84 | 80 | 84
score on a scale | 0.91 (0.23) | 2.14 (0.24) | 1.05 (0.22)
Statistical Analysis 1: Comparison: 0.75mg LY3372689 vs Placebo; Test type: Superiority; p = 0.665, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = -0.14, 95% CI 2-sided [-0.763 to 0.488], Standard Error of Mean 0.32
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Test type: Superiority; p = 0.001, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = 1.09, 95% CI 2-sided [0.435 to 1.736], Standard Error of Mean 0.33

4. Secondary Outcome: Change From Baseline to End Time Point in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) (Overall Population)
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; Total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity. LS Mean change from baseline was calculated using natural cubic spline with 2 degrees of freedom (NCS2) adjusted for fixed effects of NCS basis expansion terms (two terms), NCS basis expansion term-by-treatment interaction, visit (in weeks), investigator site (pooled), age at baseline, baseline tau PET category, AChEI/Memantine use at baseline.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline or post-baseline data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.75mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 106 | 101 | 106
score on a scale | 1.54 (0.25) | 2.81 (0.27) | 1.48 (0.25)
Statistical Analysis 1: Comparison: 0.75mg LY3372689 vs Placebo; Test type: Superiority; p = 0.878, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = 0.05, 95% CI 2-sided [-0.641 to 0.749], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Test type: Superiority; p < 0.001, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = 1.33, 95% CI 2-sided [0.615 to 2.050], Standard Error of Mean 0.36

5. Secondary Outcome: Change From Baseline to End Time Point in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13) (Intermediate (Low-medium) Tau Population)
Description: The ADAS-Cog13 is a rater administered instrument that was designed to assess the severity of the dysfunction in the cognitive and noncognitive behaviours characteristic of persons with AD. The cognitive subscale of the ADAS-Cog13 consists of 13 items assessing areas of cognitive function most typically impaired in AD: orientation, verbal memory, language, praxis, delayed free recall, digit cancellation. The ADAS-Cog13 scale ranges from 0 to 85. Higher scores indicate greater disease severity. LS Mean change from baseline was calculated using natural cubic spline with 2 degrees of freedom (NCS2) adjusted for fixed effects of NCS basis expansion terms (two terms), NCS basis expansion term-by-treatment interaction, visit (in weeks), investigator site (pooled), age at baseline, AChEI/Memantine use at baseline.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline or post-baseline data for this outcome with baseline Intermediate Tau level.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.75mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 84 | 80 | 84
score on a scale | 4.00 (0.70) | 4.91 (0.76) | 5.14 (0.69)
Statistical Analysis 1: Comparison: 0.75mg LY3372689 vs Placebo; Test type: Superiority; p = 0.252, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = -1.13, 95% CI 2-sided [-3.073 to 0.811], Standard Error of Mean 0.99
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Test type: Superiority; p = 0.825, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = -0.23, 95% CI 2-sided [-2.252 to 1.797], Standard Error of Mean 1.03

6. Secondary Outcome: Change From Baseline to End Time Point in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13) (Overall Population)
Description: The ADAS-Cog13 is a rater administered instrument that was designed to assess the severity of the dysfunction in the cognitive and noncognitive behaviours characteristic of persons with AD. The cognitive subscale of the ADAS-Cog13 consists of 13 items assessing areas of cognitive function most typically impaired in AD: orientation, verbal memory, language, praxis, delayed free recall, digit cancellation. The ADAS-Cog13 scale ranges from 0 to 85. Higher scores indicate greater disease severity. LS Mean change from baseline was calculated using natural cubic spline with 2 degrees of freedom (NCS2) adjusted for fixed effects of NCS basis expansion terms (two terms), NCS basis expansion term-by-treatment interaction, visit (in weeks), investigator site (pooled), age at baseline, baseline tau PET category, AChEI/Memantine use at baseline.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline or post-baseline data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.75mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 106 | 102 | 106
score on a scale | 5.58 (0.78) | 7.61 (0.83) | 5.95 (0.76)
Statistical Analysis 1: Comparison: 0.75mg LY3372689 vs Placebo; Test type: Superiority; p = 0.733, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = -0.37, 95% CI 2-sided [-2.527 to 1.779], Standard Error of Mean 1.09
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Test type: Superiority; p = 0.143, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = 1.66, 95% CI 2-sided [-0.565 to 3.877], Standard Error of Mean 1.13

7. Secondary Outcome: Change From Baseline to End Time Point in Alzheimer's Disease Cooperative Study Instrumental Activities of Daily Living Inventory (ADCS-iADL) (Intermediate (Low-medium) Tau Population)
Description: The ADCS-iADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The ADCS-iADL measures both basic and instrumental activities (instrumental activity items 6a, 7-23) of daily living by participants. The range for the ADCS-iADL is 0-59 with higher scores reflecting better performance. LS Mean change from baseline was calculated using natural cubic spline with 2 degrees of freedom (NCS2) adjusted for fixed effects of NCS basis expansion terms (two terms), NCS basis expansion term-by-treatment interaction, visit (in weeks), investigator site (pooled), age at baseline, AChEI/Memantine use at baseline.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline or post-baseline data for this outcome with baseline Intermediate Tau level.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.75mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 83 | 79 | 82
score on a scale | -2.65 (0.72) | -5.34 (0.77) | -2.82 (0.70)
Statistical Analysis 1: Comparison: 0.75mg LY3372689 vs Placebo; Test type: Superiority; p = 0.860, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = 0.18, 95% CI 2-sided [-1.802 to 2.158], Standard Error of Mean 1.00
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Test type: Superiority; p = 0.017, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = -2.51, 95% CI 2-sided [-4.567 to -0.456], Standard Error of Mean 1.04

8. Secondary Outcome: Change From Baseline to End Time Point in Alzheimer's Disease Cooperative Study Instrumental Activities of Daily Living Inventory (ADCS-iADL) (Overall Population)
Description: The ADCS-iADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The ADCS-iADL measures both basic and instrumental activities (instrumental activity items 6a, 7-23) of daily living by participants. The range for the ADCS-iADL is 0-59 with higher scores reflecting better performance. LS Mean change from baseline was calculated using natural cubic spline with 2 degrees of freedom (NCS2) adjusted for fixed effects of NCS basis expansion terms (two terms), NCS basis expansion term-by-treatment interaction, visit (in weeks), investigator site (pooled), age at baseline, baseline tau PET category, AChEI/Memantine use at baseline.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline or post-baseline data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.75mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 105 | 101 | 104
score on a scale | -4.02 (0.79) | -7.26 (0.83) | -3.24 (0.77)
Statistical Analysis 1: Comparison: 0.75mg LY3372689 vs Placebo; Test type: Superiority; p = 0.479, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = -0.78, 95% CI 2-sided [-2.949 to 1.387], Standard Error of Mean 1.10
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Test type: Superiority; p < 0.001, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = -4.01, 95% CI 2-sided [-6.239 to -1.788], Standard Error of Mean 1.13

9. Secondary Outcome: Change From Baseline to End Time Point in Mini Mental State Examination (MMSE) (Intermediate (Low-medium) Tau Population)
Description: MMSE is an instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures). Total score ranges from 0 to 30; lower score indicates greater disease severity. LS Mean change from baseline was calculated using natural cubic spline with 2 degrees of freedom (NCS2) adjusted for fixed effects of NCS basis expansion terms (two terms), NCS basis expansion term-by-treatment interaction, visit (in weeks), investigator site (pooled), age at baseline, AChEI/Memantine use at baseline.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline or post-baseline data for this outcome with baseline Intermediate Tau level.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.75mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 84 | 80 | 84
score on a scale | -1.65 (0.38) | -2.79 (0.41) | -2.25 (0.37)
Statistical Analysis 1: Comparison: 0.75mg LY3372689 vs Placebo; Test type: Superiority; p = 0.259, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = 0.60, 95% CI 2-sided [-0.445 to 1.642], Standard Error of Mean 0.53
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Test type: Superiority; p = 0.324, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = -0.54, 95% CI 2-sided [-1.629 to 0.541], Standard Error of Mean 0.55

10. Secondary Outcome: Change From Baseline to End Time Point in Mini Mental State Examination (MMSE) (Overall Population)
Description: MMSE is an instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures). Total score ranges from 0 to 30; lower score indicates greater disease severity. LS Mean change from baseline was calculated using natural cubic spline with 2 degrees of freedom (NCS2) adjusted for fixed effects of NCS basis expansion terms (two terms), NCS basis expansion term-by-treatment interaction, visit (in weeks), investigator site (pooled), age at baseline, baseline tau PET category, AChEI/Memantine use at baseline.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline or post-baseline data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.75mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 106 | 102 | 106
score on a scale | -2.52 (0.41) | -4.00 (0.44) | -2.70 (0.40)
Statistical Analysis 1: Comparison: 0.75mg LY3372689 vs Placebo; Test type: Superiority; p = 0.749, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = 0.18, 95% CI 2-sided [-0.946 to 1.313], Standard Error of Mean 0.57
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Test type: Superiority; p = 0.029, NCS2; A NCS model with 2 degrees of freedom (NCS2) was used; LS Mean Difference = -1.30, 95% CI 2-sided [-2.462 to -0.134], Standard Error of Mean 0.59

11. Secondary Outcome: Change From Baseline to End Time Point In Brain Tau Deposition as Measured by Flortaucipir F18 Positron Emission Tomography (PET) Scan (Intermediate (Low-medium) Tau Population)
Description: Flortaucipir PET imaging was used as a quantitative tau biomarker. Quantitative tau burden was formalized using Standardized Uptake Value Ratio (SUVR) from the following composite brain regions: frontal, parietal, occipital, and temporal lobes and the Alzheimer's disease (AD) neocortical signature. The AD neocortical signature region of interest refers to a weighted Alzheimer's Disease specific neocortical region derived from Multiblock Barycentric Discriminant Analysis. Cerebellar gray matter was used as a reference region to derive an SUVr. Larger SUVR reflects larger tau burden. LS Mean change from baseline was calculated using ANCOVA adjusted for baseline score, age and treatment (Type III sum of squares).
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline Intermediate Tau level and with baseline and at least one postbaseline PET tau data.
Measure: Least Squares Mean (Standard Error); unit: standardized uptake value ratio (SUVR)
Arm/Group | 0.75mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 68 | 57 | 70
standardized uptake value ratio (SUVR)
  Frontal | 0.05 (0.008) | 0.03 (0.009) | 0.04 (0.008)
  Parietal | 0.05 (0.009) | 0.03 (0.010) | 0.06 (0.009)
  Lateral occipital | 0.04 (0.015) | 0.05 (0.016) | 0.07 (0.015)
  Lateral temporal | 0.07 (0.011) | 0.04 (0.012) | 0.07 (0.011)
  AD neocortical signature (measured using MUBADA) | 0.07 (0.011) | 0.05 (0.012) | 0.08 (0.010)
Statistical Analysis 1: Comparison: 0.75mg LY3372689 vs Placebo; Frontal; Test type: Superiority; p = 0.346, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.01 to 0.03], Standard Error of Mean 0.012
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Frontal; Test type: Superiority; p = 0.412, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.04 to 0.01], Standard Error of Mean 0.013
Statistical Analysis 3: Comparison: 0.75mg LY3372689 vs Placebo; Parietal; Test type: Superiority; p = 0.421, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.04 to 0.02], Standard Error of Mean 0.013
Statistical Analysis 4: Comparison: 3 mg LY3372689 vs Placebo; Parietal; Test type: Superiority; p = 0.080, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.05 to 0.00], Standard Error of Mean 0.014
Statistical Analysis 5: Comparison: 0.75mg LY3372689 vs Placebo; Lateral occipital; Test type: Superiority; p = 0.192, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.07 to 0.01], Standard Error of Mean 0.021
Statistical Analysis 6: Comparison: 3 mg LY3372689 vs Placebo; Lateral occipital; Test type: Superiority; p = 0.279, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.07 to 0.02], Standard Error of Mean 0.022
Statistical Analysis 7: Comparison: 0.75mg LY3372689 vs Placebo; Lateral temporal; Test type: Superiority; p = 0.693, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.04 to 0.02], Standard Error of Mean 0.016
Statistical Analysis 8: Comparison: 3 mg LY3372689 vs Placebo; Lateral temporal; Test type: Superiority; p = 0.040, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.07 to -0.00], Standard Error of Mean 0.016
Statistical Analysis 9: Comparison: 0.75mg LY3372689 vs Placebo; AD neocortical signature (measured using MUBADA); Test type: Superiority; p = 0.838, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.03 to 0.03], Standard Error of Mean 0.015
Statistical Analysis 10: Comparison: 3 mg LY3372689 vs Placebo; AD neocortical signature (measured using MUBADA); Test type: Superiority; p = 0.055, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.06 to 0.00], Standard Error of Mean 0.016

12. Secondary Outcome: Change From Baseline to End Time Point In Brain Tau Deposition as Measured by Flortaucipir F18 Positron Emission Tomography (PET) Scan (Overall Population)
Description: Flortaucipir PET imaging was used as a quantitative tau biomarker. Quantitative tau burden was formalized using Standardized Uptake Value Ratio (SUVR) from the following composite brain regions: frontal, parietal, occipital, and temporal lobes and the Alzheimer's disease (AD) neocortical signature. The AD neocortical signature region of interest refers to a weighted Alzheimer's Disease specific neocortical region derived from Multiblock Barycentric Discriminant Analysis. Cerebellar gray matter was used as a reference region to derive an SUVr. Larger SUVR reflects larger tau burden. LS Mean change from baseline was calculated using ANCOVA adjusted for baseline score, baseline tau PET category, age and treatment (Type III sum of squares).
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline and post-baseline PET tau data.
Measure: Least Squares Mean (Standard Error); unit: SUVR
Arm/Group | 0.75mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 79 | 70 | 86
SUVR
  Frontal | 0.07 (0.011) | 0.06 (0.011) | 0.06 (0.011)
  Parietal | 0.08 (0.013) | 0.08 (0.013) | 0.07 (0.012)
  Lateral occipital | 0.08 (0.018) | 0.09 (0.018) | 0.09 (0.017)
  Lateral temporal | 0.08 (0.015) | 0.07 (0.015) | 0.08 (0.014)
  AD neocortical signature (measured using MUBADA) | 0.09 (0.014) | 0.08 (0.015) | 0.09 (0.014)
Statistical Analysis 1: Comparison: 0.75mg LY3372689 vs Placebo; Frontal; Test type: Superiority; p = 0.455, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.02 to 0.04], Standard Error of Mean 0.013
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Frontal; Test type: Superiority; p = 0.745, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.03 to 0.02], Standard Error of Mean 0.014
Statistical Analysis 3: Comparison: 0.75mg LY3372689 vs Placebo; Parietal; Test type: Superiority; p = 0.676, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.02 to 0.04], Standard Error of Mean 0.015
Statistical Analysis 4: Comparison: 3 mg LY3372689 vs Placebo; Parietal; Test type: Superiority; p = 0.794, ANCOVA; LS Mean Difference = 0.00, 95% CI 2-sided [-0.03 to 0.03], Standard Error of Mean 0.015
Statistical Analysis 5: Comparison: 0.75mg LY3372689 vs Placebo; Lateral occipital; Test type: Superiority; p = 0.643, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.05 to 0.03], Standard Error of Mean 0.021
Statistical Analysis 6: Comparison: 3 mg LY3372689 vs Placebo; Lateral occipital; Test type: Superiority; p = 0.880, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.05 to 0.04], Standard Error of Mean 0.021
Statistical Analysis 7: Comparison: 0.75mg LY3372689 vs Placebo; Lateral temporal; Test type: Superiority; p = 0.844, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.04 to 0.03], Standard Error of Mean 0.017
Statistical Analysis 8: Comparison: 3 mg LY3372689 vs Placebo; Test type: Superiority — Lateral temporal; p = 0.388, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.05 to 0.02], Standard Error of Mean 0.017
Statistical Analysis 9: Comparison: 0.75mg LY3372689 vs Placebo; AD neocortical signature (measured using MUBADA); Test type: Superiority; p = 0.815, ANCOVA; LS Mean Difference = 0.00, 95% CI 2-sided [-0.03 to 0.04], Standard Error of Mean 0.016
Statistical Analysis 10: Comparison: 3 mg LY3372689 vs Placebo; AD neocortical signature (measured using MUBADA); Test type: Superiority; p = 0.562, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.04 to 0.02], Standard Error of Mean 0.017

13. Secondary Outcome: Change From Baseline to End Time Point in Volumetric Magnetic Resonance Imaging (vMRI) Measures (Intermediate (Low-medium) Tau Population)
Description: MRI scans at baseline and at 76 weeks after the first treatment were used to quantitatively estimate change in brain atrophy. Volumetric MRI (vMRI) parameters were measured in brain regions: bilateral hippocampus, bilateral whole lateral ventricles, and bilateral whole brain. The atrophy was assessed by tensor-based morphometry, which captures volume changes within the deformation map. LS Mean change from baseline was determined by mixed model repeated measures (MMRM) model with fixed effects of treatment, visit, treatment-by-visit interaction, and adjusted for baseline volume, age at baseline.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline Intermediate Tau level and with baseline and at least one postbaseline vMRI data.
Measure: Least Squares Mean (Standard Error); unit: cubic centimeter (cm^3)
Arm/Group | 0.75mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 68 | 61 | 75
cubic centimeter (cm^3)
  Bilateral Hippocampus | -0.19 (0.017) | -0.16 (0.019) | -0.28 (0.016)
  Bilateral Whole Lateral Ventricles | 3.52 (0.425) | 4.25 (0.458) | 5.89 (0.405)
  Bilateral Whole Brain | -10.75 (1.231) | -9.56 (1.345) | -18.92 (1.186)
Statistical Analysis 1: Comparison: 0.75mg LY3372689 vs Placebo; Bilateral Hippocampus; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = 0.09, 95% CI 2-sided [0.04 to 0.14], Standard Error of Mean 0.024
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Bilateral Hippocampus; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = 0.13, 95% CI 2-sided [0.08 to 0.18], Standard Error of Mean 0.025
Statistical Analysis 3: Comparison: 0.75mg LY3372689 vs Placebo; Bilateral Whole Lateral Ventricles; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -2.37, 95% CI 2-sided [-3.53 to -1.21], Standard Error of Mean 0.587
Statistical Analysis 4: Comparison: 3 mg LY3372689 vs Placebo; Bilateral Whole Lateral Ventricles; Test type: Superiority; p = 0.008, Mixed Models Analysis; LS Mean Difference = -1.64, 95% CI 2-sided [-2.84 to -0.43], Standard Error of Mean 0.611
Statistical Analysis 5: Comparison: 0.75mg LY3372689 vs Placebo; Bilateral Whole Brain; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = 8.17, 95% CI 2-sided [4.79 to 11.56], Standard Error of Mean 1.715
Statistical Analysis 6: Comparison: 3 mg LY3372689 vs Placebo; Bilateral Whole Brain; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = 9.37, 95% CI 2-sided [5.81 to 12.92], Standard Error of Mean 1.804

14. Secondary Outcome: Change From Baseline to End Time Point in Volumetric Magnetic Resonance Imaging (vMRI) Measures (Overall Population)
Description: MRI scans at baseline and at 76 weeks after the first treatment were used to quantitatively estimate change in brain atrophy. Volumetric MRI (vMRI) parameters were measured in brain regions: bilateral hippocampus, bilateral whole lateral ventricles, and bilateral whole brain. The atrophy was assessed by tensor-based morphometry, which captures volume changes within the deformation map. LS Mean change from baseline was determined by mixed model repeated measures (MMRM) model with fixed effects of treatment, visit, treatment-by-visit interaction, and adjusted for baseline volume, baseline tau PET category, age at baseline.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline and at least one postbaseline vMRI data.
Measure: Least Squares Mean (Standard Error); unit: cm^3
Arm/Group | 0.75mg LY3372689 | 3 mg LY3372689 | Placebo
Number analyzed (Participants) | 82 | 78 | 94
cm^3
  Bilateral Hippocampus | -0.21 (0.018) | -0.17 (0.018) | -0.29 (0.017)
  Bilateral Whole Lateral Ventricles | 4.95 (0.444) | 5.74 (0.455) | 7.16 (0.409)
  Bilateral Whole Brain | -15.61 (1.292) | -14.62 (1.313) | -22.78 (1.195)
Statistical Analysis 1: Comparison: 0.75mg LY3372689 vs Placebo; Bilateral Hippocampus; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = 0.08, 95% CI 2-sided [0.04 to 0.13], Standard Error of Mean 0.023
Statistical Analysis 2: Comparison: 3 mg LY3372689 vs Placebo; Test type: Superiority — Bilateral Hippocampus; p < 0.001, Mixed Models Analysis; LS Mean Difference = 0.12, 95% CI 2-sided [0.08 to 0.17], Standard Error of Mean 0.023
Statistical Analysis 3: Comparison: 0.75mg LY3372689 vs Placebo; Bilateral Whole Lateral Ventricles; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -2.21, 95% CI 2-sided [-3.33 to -1.08], Standard Error of Mean 0.570
Statistical Analysis 4: Comparison: 3 mg LY3372689 vs Placebo; Bilateral Whole Lateral Ventricles; Test type: Superiority; p = 0.015, Mixed Models Analysis; LS Mean Difference = -1.42, 95% CI 2-sided [-2.57 to -0.28], Standard Error of Mean 0.582
Statistical Analysis 5: Comparison: 0.75mg LY3372689 vs Placebo; Bilateral Whole Brain; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = 7.17, 95% CI 2-sided [3.95 to 10.40], Standard Error of Mean 1.635
Statistical Analysis 6: Comparison: 3 mg LY3372689 vs Placebo; Bilateral Whole Brain; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = 8.16, 95% CI 2-sided [4.85 to 11.47], Standard Error of Mean 1.680

15. Secondary Outcome: Pharmacokinetics (PK): Plasma Concentrations of LY3372689
Description: Blood samples were measured at week 64 to assess the concentration of LY3372689 in the plasma.
Time Frame: Week 64: Post-dose
Population: All randomized participants who received at least one 1 of study drug and had evaluable C-trough data at the specified time points
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 0.75 mg LY3372689 | 3 mg LY3372689
Number analyzed (Participants) | 76 | 69
nanograms per milliliter (ng/mL) | 3.95 (163) | 12.9 (212)

ADVERSE EVENTS:
Time Frame: Baseline Up To 124 Weeks
Description: All randomized participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had number of participants at risk adjusted accordingly.
  One death is noted in participant flow for '3 mg LY3372689' arm, while two are reported under adverse events. This is because a participant who discontinued due to an AE later died-counted as "AE leading to death" in adverse events, but only as "discontinuation due to AE" in participant flow.
Arm/Group | 0.75mg LY3372689 | 3 mg LY3372689 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/108 | 2/110 | 1/108
Serious Adverse Events (participants affected / at risk) | 13/108 | 29/110 | 17/108
Other Adverse Events (participants affected / at risk) | 74/108 | 72/110 | 81/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.75mg LY3372689 (N=108) | 3 mg LY3372689 (N=110) | Placebo (N=108)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dental sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative delirium (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haematological malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dementia of the alzheimer's type, with delirium (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 0.75mg LY3372689 (N=108) | 3 mg LY3372689 (N=110) | Placebo (N=108)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 6 (6) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 13 (18) | 12 (17) | 12 (14)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8) | 8 (11) | 7 (8)
Fatigue (General disorders) | 2 (2) | 6 (6) | 5 (5)
Covid-19 (Infections and infestations) | 24 (27) | 17 (18) | 23 (24)
Nasopharyngitis (Infections and infestations) | 5 (5) | 7 (8) | 9 (10)
Upper respiratory tract infection (Infections and infestations) | 14 (17) | 11 (13) | 8 (8)
Urinary tract infection (Infections and infestations) | 8 (11) | 8 (13) | 13 (21)
Fall (Injury, poisoning and procedural complications) | 20 (27) | 16 (37) | 15 (19)
Electrocardiogram pr prolongation (Investigations) | 4 (10) | 8 (15) | 5 (6)
Electrocardiogram qt prolonged (Investigations) | 8 (15) | 10 (16) | 5 (10)
Weight decreased (Investigations) | 6 (6) | 8 (9) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 4 (5) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 5 (5) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2) | 6 (6)
Dizziness (Nervous system disorders) | 7 (9) | 8 (13) | 9 (9)
Headache (Nervous system disorders) | 16 (88) | 13 (15) | 6 (6)
Tremor (Nervous system disorders) | 4 (4) | 6 (8) | 2 (2)
Anxiety (Psychiatric disorders) | 8 (9) | 8 (8) | 5 (9)
Depression (Psychiatric disorders) | 7 (8) | 2 (2) | 3 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2/39 (2) | 2/46 (2) | 0/40 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 3 (3) | 6 (8)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT05063539/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT05063539/SAP_001.pdf